CLINICAL TRIAL: NCT06663995
Title: Evaluation of Locally Delivered Propolis Gel As an Adjunct to Nonsurgical Periodontal Therapy in the Management of Periodontitis: a Randomized Controlled Clinical Study with Biochemical Assessment
Brief Title: Evaluation of Locally Delivered Propolis Gels in Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Huda Mohamed, BDS, Clinical demonstrator, oral medicine and periodontology, Horus University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RecIM122223
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SRP (Placebo Comparator): The participants were randomly assigned to receive medicated with SRP combined with intrasulcular application of placebo gel. After baseline assessment, at the same day the included participants will receive full mouth one stage debridement using hand instruments and ultrasonic scalers under local anesthesia -if needed- for patient's comfort. Participants will be provided with a toothpaste, a medium toothbrush, a written oral hygiene instruction brochure (Brushing twice daily for 4-weeks using Modified Bass technique and interdental flossing).
  Interventions: Drug: Control (placebo) group
- PROPOLIS group (Active Comparator): After baseline assessment, at the same day the included participants will receive full mouth one stage debridement using hand instruments and ultrasonic scalers under local anesthesia -if needed- for patient's comfort.
  2- Oral Hygiene Instructions Participants will be provided with a toothpaste, a medium toothbrush, a written oral hygiene instruction brochure (Brushing twice daily for 4-weeks using Modified Bass technique and interdental flossing).
  3-Base line visit (Local delivery application): Propolis gel will be applied by syringe with blunt tip gently and removed slowly in order not to harm the tissue for group 1 patients (Test group) after phase 1 therapy at the second day (48 hours) following non-surgical periodontal therapy
  Interventions: Drug: Study Group

INTERVENTIONS:
Drug: Study Group — It will include 16 patients with periodontitis stage II, grade B, at least 2 sites with pocket PD = 4-5 mm and CAL = 3-4 mm each will receive non-surgical periodontal therapy followed by application of propolis gel.
  After baseline assessment, at the same day the included participants will receive full mouth one stage debridement using hand instruments and ultrasonic scalers under local anesthesia -if needed- for patient's comfort.
  2- Oral Hygiene Instructions Participants will be provided with a toothpaste, a medium toothbrush, a written oral hygiene instruction brochure (Brushing twice daily for 4-weeks using Modified Bass technique and interdental flossing).
  3-Base line visit (Local delivery application): Propolis gel will be applied by syringe with blunt tip gently and removed slowly in order not to harm the tissue for group 1 patients (Test group) after phase 1 therapy at the second day (48 hours) following non-surgical periodontal therapy
  Arms: PROPOLIS group
Drug: Control (placebo) group — After baseline assessment, at the same day the included participants will receive full mouth one stage debridement using hand instruments and ultrasonic scalers under local anesthesia -if needed- for patient's comfort.
  2- Oral Hygiene Instructions Participants will be provided with a toothpaste, a medium toothbrush, a written oral hygiene instruction brochure (Brushing twice daily for 4-weeks using Modified Bass technique and interdental flossing).
  Arms: SRP

SUMMARY:
Assess the efficacy of locally delivered propolis gel as an adjunct to scaling and root planning in management of Stage II, Grade B periodontitis

. Subjects and Methods

I. Patients' selection:

Thirty-two (32) patients were recruited from the outpatient clinic of Oral Medicine, Periodontology, and Oral Diagnosis department, Faculty of Dentistry, Ain Shams University.

This study was designed as a randomized, controlled, 2-parallel arm, triple blinded, single center clinical trial.

Thirty-two eligible patients with stage II and Grade B periodontitis were randomly assigned into 2 groups:

* Group 1 (intervention group) was treated with SRP combined with intrasulcular application of 1% Propolis gel.
* Group 2 (control group) was treated with SRP combined with intrasulcular application of placebo gel.

DETAILED DESCRIPTION:
Thirty-two eligible patients with stage II and Grade B periodontitis were randomly assigned into 2 groups:

* Group 1 (intervention group) was treated with SRP combined with intrasulcular application of 1% Propolis gel.
* Group 2 (control group) was treated with SRP combined with intrasulcular application of placebo gel.

Eligibility criteria:

The patients were recruited according to the following criteria:

Inclusion criteria

1. Both genders aged from 30-50 years
2. Systemically healthy patients were classified as ASA class I, II as evidenced by (modified Cornell medical index)
3. Patients with Stage II, Grade B Periodontitis, according to the 2017 world workshop on the classification of periodontal and peri- implant disease and conditions. Interdental CAL at site of greatest depth 3-4 mm, bleeding on probing (BOP), maximum PD ≤5mm and radiographic horizontal bone loss related to the coronal third of the root (15%-33%), with no history of periodontal therapy or use of antibiotics in the preceding 6 months
4. Patient with no history of periodontal therapy or use of antibiotics or anti-inflammatory in the preceding 6 months.
5. Patient willing to comply with oral hygiene instructions. Exclusion criteria

<!-- -->

1. Patients with known allergy to propolis.
2. Smokers or Alcoholics patients.
3. Pregnant and lactating females

Study Design, Randomization and Blinding:

This study was designed as a randomized, controlled, 2-parallel arm, triple blinded, single center clinical trial.

Thirty-two eligible patients with stage II and Grade B periodontitis were randomly assigned into 2 groups:

* Group 1 (intervention group) was treated with SRP combined with intrasulcular application of 1% Propolis gel.
* Group 2 (control group) was treated with SRP combined with intrasulcular application of placebo gel.

The participants were randomly assigned to receive medicated formula of Propolis or Placebo using a randomization procedure with a 1:1 allocation ratio. A computer-generated randomization list using randomizer.org website was executed by the co-supervisor who was not involved in the recruitment for the purpose of concealment Allocation concealment was achieved by co-supervisor (D. A.) who had the randomization list, and was contacted by phone after confirming the eligibility of the participant to be allocated to either Propolis group or Placebo group according to the random sequence known by the co- supervisor.

The current trial was a triple-blinded clinical trial. Blinding included patients, principal investigator and the outcome assessors.

Patients who met the eligibility criteria were assessed clinically for the following clinical parameters using the University of North Carolina probe (UNC15)1 (Figure 2). The clinical parameters were recorded in the online colored periodontal chart by the Periodontology Department, University of Bern 20102 (

Interventions:

Propolis and placebo Gel Preparation

* 100 ml of Placebo gel was prepared by mixing 3.344 g of carboxymethylcellulose sodium salt (CMC; El Nasr Pharmaceutical Chemicals Co., Egypt).
* 200 mg methyl hydroxy benzoate sodium salt (Loba Chemie, India) as a preservative in 81.77 mL of double distilled water (dDW).
* 18.22 ml of HPLC-grade ethanol (Merck, Germany) under continuous stirring overnight to ensure complete solubilization of the CMC.
* To prepare 100 ml of propolis extract gel, 1 g of propolis (Imtnan, Egypt) was extracted using 18.22 ml ethanol.
* then 10 g of propylene glycol was added to the ethanolic extract to enhance its solubility in the aqueous phase.
* The propolis gel was then prepared by the same method as that of the placebo gel by adding 3.344 g of CMC dissolved in water to the above mixture and completing the total weight to 100 g using distilled water .

The gel was filled in 20 syringes (5ml) and kept in the refrigerator.

Treatment Protocol:

1. Phase I periodontal therapy and periodontal charting:

   * Initial examination was done including full mouth probing using UNC15 Periodontal probe followed by periapical radiographic examination for the selected sites (PPD ≤5mm).
   * Patient motivation and education for proper oral hygiene instructions included twice-daily tooth brushing with soft toothbrush using modified bass brushing technique and once daily interdental cleaning with dental floss and interdental brushes for wide interproximal embrasure spaces.
   * Full mouth supra and subgingival debridement was performed using ultrasonic device4 with supragingival scaling tips followed by universal and Gracey's curettes 5 for proper subgingival debridement. Local anesthesia6 was used for patient's comfort whenever needed.
   * After 48 hours from the last periodontal instrumentation visit, patients were recalled for recording baseline clinical parameters and collecting the baseline GCF sample, then local drug application.
2. Gingival crevicular fluid Sampling:

Gingival crevicular fluid (GCF) samples were collected from Thirty-two (32) selected sites, one in each patient; selected sites were isolated using cotton rolls and gently dried. A standard paper strip7 was inserted into the sulcus until resistance is felt for 30 seconds and then removed, after collection of gingival fluid the strips were placed in sterile Eppendorf tubes containing 100 ul phosphate buffer PH 7.4 and stored at -20 o C till time of analysis.

GCF samples were stored at -20 C until further analysis after collecting all the samples in baseline,1 month and 3 months duration for all patients for biological assessment.

1- interventions:

After collecting GCF samples, application of the interventions takes place; either Propolis or Placebo according to the random sequence.

A sterile 1ml micro-syringe9 was filled with the medication and then it was injected using plastic tip into the sulcus, filling the whole interdental area

1- Clinical parameters:

All clinical periodontal parameters were assessed at baseline, after 3 months and 6 months.

The following parameters were assessed preoperatively:

1. Clinical attachment level (CAL).(Ramfjord 1967)
2. Probing depth (PD). (Listgarten 1980)
3. Gingival index (GI) (Löe 1967)).
4. Plaque index (PI). (Loe 1964)

<!-- -->

1. Clinical attachment level (CAL) (Ramfjord, 1967):

   CAL was measured as the distance between the fixed reference points, i.e., CEJ to the base of the pocket and recorded manually for six sites at each tooth.

   o Two parameters were recorded concerning CAL:

   - Mean CAL: CAL was measured for each patient (total CAL at all sites/number of surfaces).

   - Mean Highest CAL site: The highest clinical attachment loss measure for each patient was recorded and the mean of highest CAL was calculated for each group, and this was considered as the primary outcome
2. Periodontal pocket depth (PPD) (Listgarten, 1980):

   In order to measure PPD, the probe was inserted parallel to the long axis of the tooth to reach the deepest point of the pocket, and the distance between the base of the pocket and gingival margin was recorded manually to the nearest millimeter marking. Six readings were recorded for each tooth.

   o Two parameters were recorded concerning PPD:

   - Mean PPD: The PPD was measured for each patient (total PD/number of surfaces).

   - Mean Deepest PPD: The deepest pocket measure for each patient was recorded and the mean of deepest pocket was calculated for each group.
3. Gingival index (GI) (Löe 1967)):

   The gingival criteria were assessed using the following score:

   • 0 = normal gingival.

   • 1 = mild inflammation: slight change in color, slight edema, no bleeding on probing.

   • 2 = moderate inflammation: redness, edema, and glazing, or bleeding on probing.
   * 3 = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding, ulceration.

     * GI was measured on two surfaces of teeth (buccal and lingual) and a mean was taken for all teeth and recorded for each patient.
4. Plaque index (PI) (Loe 1964)):

The plaque deposits on the surface of teeth were assessed and scored as following:

* 0=No plaque
* 1= A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
* 2= Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
* 3= Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.

  * PI was measured on two surfaces of teeth (buccal and lingual) and a mean was taken for all teeth and recorded for each patient

Quantitative biomechanical assessment:

The examined area will be dried by gentle air stream and isolated with cotton rolls to prevent contamination with saliva. Next, with sterile tweezers one perio paper will be inserted into the selected pocket and left in situ for 30 seconds. Perio paper are placed in sterile Eppendorf tubes containing 100 ul phosphate buffer PH 7.4 and stored at -20 o C till time of analysis.

Samples will be analyzed to assess the level of prostaglandin E2 (PGE2) by using commercially available ELISA kits by following the instructions of the manufacturer. For all patients, Gingival crevicular fluid (GCF) samples will be taken and analyzed at baseline and three months after periodontal treatment .

ELIGIBILITY:
Inclusion Criteria:

* 1-Both genders aged from 30-50 years 2- Systemically healthy patients as evidenced by (modified Cornell medical index) (Pendleton et al., 2004).

  3- Patients with Stage II, Grade B Periodontitis, Test sites at least 2 sites have Propping depth (PD)= 4-5 mm or Clinical attachment loss (CAL)= 3-4mm.

  4- Patient with no history of periodontal therapy or use of antibiotics or anti-inflammatory in the preceding 6 months.

  5- Patient willing to comply with oral hygiene instructions

Exclusion Criteria:

* 1-Patients with known allergy to propolis. 2- Smokers or Alcoholics patients. 3- Pregnant and lactating females.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-17 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Regarding clinical periodontal parameters as a primary objective. | The following clinical parameters will be recorded for the individuals preoperatively and 3 and 6 months postoperatively.
  Probing pocket depth will be measured from the gingival margin to the base of the periodontal pocket to the nearest mm. with use of periodontal probe.

SECONDARY OUTCOMES:
B) Secondary outcome: • Biochemically By analyzing quantitative changes the level of prostaglandin E2 (PGE2) in the gingival crevicular fluid (GCF) | The examined area will be dried by gentle air stream and isolated with cotton rolls to prevent contamination with saliva. Next, with sterile tweezers one perio paper will be inserted into the selected pocket and left in situ for 30 seconds. Perio paper a

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided